CLINICAL TRIAL: NCT03707210
Title: Virtual Reality Application in Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N201902009; N201902009 (Registry Identifier: TMU-JIRB)
Record Dates: First submitted 2018-10-02; First posted 2018-10-16 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2018-07

CONDITIONS: Chemotherapy Training
Keywords: virtual reality; chemotherapy

STUDY DESIGN:
Intervention Model Description: intervention: VR training; control group: ISO document
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group uses the VR program to training chemotherapy skill. Use VR software to make a training education program.
  Interventions: Behavioral: VR training program
- usual care (No Intervention): Chemotherapy training as usual care (for training chemotherapy skill).

INTERVENTIONS:
Behavioral: VR training program — Use VR software to make a training education program.
  Arms: Intervention

SUMMARY:
The present study wants to design a training program for chemotherapy with using VR. Then the investigators design a protocol to compare the training effects in the VR program and ISO document.

DETAILED DESCRIPTION:
As technology advances, mobile devices have gradually turned into wearable devices. Furthermore, virtual reality (VR), augmented reality (AR), and mixed reality (MR) are being increasingly applied in medical fields such as medical education and training, surgical simulation, neurological rehabilitation, psychotherapy, and telemedicine. Research results demonstrate the ability of VR, AR, and MR to ameliorate the inconveniences that are often associated with traditional medical care, reduce incidents of medical malpractice caused by unskilled operations, and reduce the cost of medical education and training. What is more, the application of these technologies has enhanced the effectiveness of medical education and training, raised the level of diagnosis and treatment, improved the doctor-patient relationship, and boosted the efficiency of medical execution. The present study wants to design a training program for chemotherapy with using VR. Then the investigators design a protocol to compare the training effects in VR program and ISO document.

ELIGIBILITY:
Inclusion Criteria:

1. The staffs who require to implement chemotherapy skill in the hospital.
2. Age over 20 years.

Exclusion Criteria:

1. Refuse to join the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
The questionnaire about intervention effect | After intervention 1 week, to perform the test. Including the content design, the convenience, the effectiveness, and promotion.
  After intervention, the investigator want to know the effect of intervention. A total of 12 questions, using the Likert's scale, very disagree(1) to very agree(5). It will compute a total score, score high means more effective.

SECONDARY OUTCOMES:
The questionnaire of Knowledge level for chemotherapy technique | Before the intervention, the investigator perform a pretest. After intervention 1 week, the investigator perform the post test.
  The questionnaire want to understand the Knowledge for chemotherapy operation skill before and after intervention. A total of ten questions, with scores ranging from 0 to 10 points. , score high means more correct.
The questionnaire of Attitude for chemotherapy operation | Before the intervention, the investigator perform a pretest. After intervention 1 week, the investigator perform the post test.
  The questionnaire want to understand the Attitude for chemotherapy operation skill before and after intervention. A total of ten questions, using the likert's scale, very disagree with 1 point, very agree with 5 points, total scores between 10 points and 50 points. , score high means more active.

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Wei Huang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Chan HY, Chang HC, Huang TW. Virtual reality teaching in chemotherapy administration: Randomised controlled trial. J Clin Nurs. 2021 Jul;30(13-14):1874-1883. doi: 10.1111/jocn.15701. Epub 2021 Feb 18. PMID 33555626